CLINICAL TRIAL: NCT06976437
Title: An Exploratory Clinical Study on the Safety and Efficacy of Allogeneic CD19/BCMA CAR-T Cell Treatment for Relapsed/ Refractory B-cell or Plasma Cell-derived Malignant Tumors
Brief Title: A Clinical Study of Allogeneic CD19/BCMA CAR-T Cells for the Treatment of R/R B-cell Malignant Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: YANRU WANG (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry); Allorunning Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, YANRU WANG, Doctor, Affiliated Hospital of Jiangsu University
Organization: Affiliated Hospital of Jiangsu University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RunNing
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: B Cell Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, B-Cell; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RN1101 treatment (Experimental): CD19+ or BCMA+ r/r B Cell lymphoma or multiple myeloma (MM) patients to be treated with a single dose of RN1101 cells.
  Interventions: Drug: RN1101 injection

INTERVENTIONS:
Drug: RN1101 injection — RN1101 injection is an allogenic CAR-T targeted CD19 and BCMA. A single infusion of CAR-T cells will be administered intravenously.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and efficacy of CD19 and B-cell maturation antigen (BCMA) targeted allogenic CAR-T cells (RN1101) in patients with relapsed/refractory B-cell or plasma cell-derived malignant tumors. 21 patients are planned to be enrolled in the dose-escalation trial. The primary objective of the study is to evaluation of the safety and feasibility of RN1101 for the treatment of relapsed/refractory B-cell or plasma cell-derived malignant tumors. The secondary objective is to evaluate the efficacy of RN1101 for the treatment of relapsed/refractory B-cell or plasma cell-derived malignant tumors. The exploratory objective is to evaluate expansion, persistence and ability of RN1101 to deplete CD19 or BCMA positive cells in patients with relapsed/refractory B-cell or plasma cell-derived malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to participate in the trial and provision of signed informed consent.
2. Patients diagnosed with B-lymphocyte or plasma cell-derived malignancies as per the 2017 revised WHO criteria, including acute B-lymphoblastic leukemia (B-ALL), and mature B-cell lymphomas such as diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), marginal zone lymphoma (MZL), small lymphocytic lymphoma/chronic lymphocytic leukemia (SLL/CLL), mantle cell lymphoma (MCL), multiple myeloma (MM), etc.
3. Refractory or recurrent B-lymphocyte or plasma cell-derived malignancies, defined as failure to achieve complete remission after standard treatment, or relapse during follow-up after achieving remission with first-line or salvage therapy.
4. Patients with B-cell acute lymphoblastic leukemia (ALL) who have achieved hematologic remission but have persistent minimal residual disease (MRD).
5. According to the revised International Working Group (IWG) criteria, relapsed/refractory lymphoma patients must have at least one measurable lesion with a longest diameter ≥1.5 cm.
6. 18 Years and older, regardless of gender.
7. An expected survival of ≥12 weeks.
8. Serum total bilirubin level < twice the upper limit of normal, serum creatinine level < upper limit of normal, serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < three times the upper limit of normal.
9. Absolute neutrophil count ≥0.5×10⁹/L, platelets ≥20×10⁹/L; for B-lymphocyte malignancies with definitive bone marrow involvement, no requirements for neutrophil and platelet counts.
10. ECOG performance status of 0 - 2.
11. Left ventricular ejection fraction (LVEF) ≥50% and no pericardial effusion.
12. At least 2 weeks have passed since the last treatment (radiotherapy, chemotherapy, monoclonal antibody therapy, or other treatments).

Exclusion Criteria:

1. Known allergies, hypersensitivity, intolerance, or contraindications to CD19/BCMA allogenic CAR-T or any components of the trial drugs (including fludarabine, cyclophosphamide, and rituximab), or a history of severe allergic reactions.
2. Recurrence after allogeneic hematopoietic stem cell transplantation with active graft - versus - host disease (GVHD) requiring steroid or immunosuppressive therapy.
3. Severe active infection.
4. Acquired or congenital immunodeficiency.
5. New York Heart Association (NYHA) Class Ⅲ or Ⅳ heart failure.
6. History of epilepsy or other central nervous system diseases.
7. Lymphoma with extranodal involvement of the brain, lungs, or gastrointestinal tract.
8. Other primary cancers, except:

   1. Non-melanoma skin cancer (e.g., basal cell carcinoma) cured by resection.
   2. Carcinoma in situ (e.g., cervical, bladder, or breast cancer) cured.
9. Systemic high-dose steroids within 2 weeks before treatment.
10. Pregnant, breastfeeding, or plans to become pregnant within 6 months.
11. Participation in another clinical trial within the past month.
12. Any situation the investigator deems may raise risks or interfere with trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events after RN1101 infusion | up to 24 weeks after RN1101 infusion

SECONDARY OUTCOMES:
Percentage of MRD negative patients after RN1101 treatment | 12 weeks, 24 weeks after RN1101 infusion
ORR (PR, VGPR, CR and sCR) of patients receive RN1101 treatment | 12 weeks, 24 weeks after RN1101 infusion
Progression free survival after RN1101 treatment | 12 weeks, 24 weeks after RN1101 infusion
CAR copies and cell count of CAR-T in blood and bone marrow (if available) after RN1101 treatment | 12 weeks, 24 weeks after RN1101 infusion
Duration of response after RN1101 treatment | 12 weeks, 24 weeks after RN1101 infusion
Overall survival after RN1101 treatment | 12 weeks, 24 weeks after RN1101 infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No